CLINICAL TRIAL: NCT01354782
Title: An Open, Single Centre, Single and Repeated Dose Study to Investigate the Pharmacokinetic Profile of Roflumilast and Roflumilast N-oxide After Administration of 500 μg Dose of Roflumilast in Healthy Chinese Subjects
Brief Title: Pharmacokinetic Study of Single and Repeated Dose of Roflumilast 500 µg , in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RO-2455-101-EC
Record Dates: First submitted 2011-05-16; First posted 2011-05-17 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Pharmacokinetic; Roflumilast
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Roflumilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Roflumilast (Experimental): (This is a pharmacokinetic study)
  Interventions: Drug: Roflumilast

INTERVENTIONS:
Drug: Roflumilast — Period I: single dose of roflumilast 500 μg orally in the morning.
  Period II: repeated dose of roflumilast 500 μg orally in the morning for 14 days.

SUMMARY:
The primary objective is to assess the pharmacokinetics (PK) of roflumilast and its metabolite roflumilast N-oxide after single and repeated oral administrations of roflumilast 500 μg in healthy Chinese subjects.

ELIGIBILITY:
Main Inclusion Criteria:

* Healthy male and female (24 male and 8 female) subjects of Chinese ethnic origin, age 40 years and older.
* Assessed as healthy based on a screening examination including medical history, physical examination, blood pressure, pulse rate, ECG assessment, and clinical laboratory results.
* Body weight according to a Body Mass Index (BMI) between 19 and 28 kg/[m²], (both inclusive) and a body weight ≥ 50 kg.
* Females with childbearing potential who are using medically acceptable and reliable method of contraception for the entire study duration, such as tubal ligation, hysterectomy, intrauterine device without hormones or post-menopausal females, the latter is defined as females who have had no menstrual period for at least 2 years.

Main Exclusion Criteria:

* History or current evidence of clinically relevant allergies or idiosyncrasy to drugs or food
* History of allergic reactions to roflumilast or any inactive ingredients of the trial medication
* History or current evidence of any clinically relevant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, hematological, endocrinological, metabolic, neurological, psychiatric, or other disease (within the last 2 years)
* History of malignancy within the past 5 years
* Electrocardiogram (ECG) abnormalities of clinical relevance (e.g. QTc according to Bazett's formula: QTc > 450 msec (male), QTc > 470 msec (female), PQ ≥ 220 msec)
* Blood pressure ≥ 140 mm HG systolic or ≥ 90 mm HG diastolic
* Elevated transaminases > 2 x upper Limit of normal range and or increased of the total bilirubin > 1.5 upper Limit of normal range
* Clinically relevant abnormalities in clinical chemical, hematological or any other laboratory variables
* Chronic or clinically relevant acute infections
* Proneness to orthostatic dysregulation, faintings, or blackouts
* Positive results in any of the virology tests of acute or chronic infectious HIV and hepatitis A, B, and C virus infections
* Positive drug screen
* Abuse of alcohol or drugs
* Positive β-HCG pregnancy test (female)
* Pregnant or lactating females

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-05; Primary Completion 2011-06 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
To determine the pharmacokinetic profiles after single and repeated dose of roflumilast 500 µg administered to healthy Chinese subjects. | Period I: single dose, PK-Investigation over 8 days, Period II: repeated dose for 14 days, PK-Investigation on days 14 and 15
  PK samples at pre-dose, 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 5h, 6h, 8h, 10h, 12h, 16h and 24h, 36h, 48h, 72h, 96h, 120h, 144h and 168h post dose after single dose and at the time points pre-dose, 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 5h, 6h, 8h, 10h, 12h, 16h and 24h after administration of a repeated dose

SECONDARY OUTCOMES:
The safety and tolerability of single and repeated dose roflumilast 500 µg will be evaluated in terms of adverse event, ECG, blood pressure, pulse rate, and clinical laboratory tests. | During screening, clinical part and final check

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (1):
- Nycomed Investigational Site, Beijing, China

REFERENCES:
- See also: RO-2455-101-EC-RDS-2012-04-26.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4497&filename=RO-2455-101-EC-RDS-2012-04-26.pdf